CLINICAL TRIAL: NCT01228019
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy Profile of TREDAPTIVE Tablet in Usual Practice
Brief Title: Niacin (+) Laropiprant (TREDAPTIVE) Re-examination Study (MK-0524A-119)
Status: Terminated | Type: Observational
Why Stopped: In HPS2-THRIVE, MK-0524A did not meet the primary efficacy objective and there was a significant increase in incidence of some types of non-fatal SAEs
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0524A-119
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Usual practice re-examination
MeSH Terms: conditions — Hypercholesterolemia | interventions — Niacin; MK-0524

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Participants with primary hypercholesterolemia or mixed dyslipidemia treated with niacin (+) laropiprant (TREDAPTIVE)
  Interventions: Drug: Niacin (+) laropiprant

INTERVENTIONS:
Drug: Niacin (+) laropiprant — Niacin (+) laropiprant (TREDAPTIVE) prescribed according to the current local label
  Other Names: MK-0524A

SUMMARY:
This survey is being conducted to assess the safety and efficacy of niacin (+) laropiprant (TREDAPTIVE) in usual practice in Korea according to the new product re-examination regulations of the Korean Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are treated with TREDAPTIVE tablet within current local label for the first time
* Participants with primary hypercholesterolemia or mixed dyslipidemia
* Participants who are treated with TREDAPTIVE for more than or equal to 24 weeks will be included in long-term surveillance
* Special participants with known hepatic disorder or renal disorder, participants 65 years old or older, participants younger than 19 years old, and pregnant woman will be evaluated if collected.

Exclusion Criteria:

* Participant who is treated with TREDAPTIVE tablet before contract and out of enrollment period
* Participant who has a contraindication to TREDAPTIVE tablet according to the current local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean participants with hypercholesterolemia or mixed dyslipidemia treated with niacin (+) laropiprant (TREDAPTIVE) for the first time
Sampling Method: Probability Sample
Enrollment: 1166 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,166 participants who were currently using niacin (+) laropiprant (TREDAPTIVE) for treatment of primary hypercholesterolemia or mixed dyslipidemia were enrolled and their case report forms were collected. Enrollment was stopped early due to termination of all studies involving TREDAPTIVE.
Pre-assignment Details: A completer was considered a participant eligible for safety population. Efficacy population was a sub-population of the safety population
Period: Overall Study
Arm/Group | All Participants
Started | 1166
Completed | 862
Not Completed | 304
Not completed — Dose Violation | 70
Not completed — Duplicate enrollment | 1
Not completed — Missing pre-treatment data | 72
Not completed — Triglyceride Entry Criteria Not Met | 152
Not completed — Violation of Entry Criterion | 9

BASELINE CHARACTERISTICS:
Population: Baseline characteristics presented for participants in the Safety Population
Arm/Group | All Participants
Number analyzed (Participants) | 862
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.03 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268
  Male | 594

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Experience
Description: An adverse event was any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the study drug, was also an adverse event.
Time Frame: From start of treatment through 14 days after the last dose (Up to 26 weeks)
Population: Safety population: all enrolled participants who met entry criteria regarding safety data
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 862
Percentage of participants | 19.61

2. Primary Outcome: Percentage of Participants With Adverse Drug Reactions
Description: An adverse drug reaction was an adverse event of which the relationship to the study drug could not be ruled out. An adverse event was any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the study drug, was also an adverse event.
Time Frame: From start of treatment through 14 days after the last dose (Up to 26 weeks)
Population: Safety population: all enrolled participants who met entry criteria regarding safety data
Measure: Number; unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 862
Percentage of Participants | 15.20

3. Primary Outcome: Change From Baseline in Total Cholesterol at Week 12
Description: Serum cholesterol levels were measured at start of treatment (baseline) and after 12 weeks of treatment with TREDAPTIVE
Time Frame: Baseline and Week 12
Population: Participants in safety population whose case report form contained baseline and Week 12 data for total cholesterol levels.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 301
mg/dL | -12.52 (32.44)

4. Primary Outcome: Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: Serum LDL-C levels were measured at start of treatment (baseline) and after 12 weeks of treatment with TREDAPTIVE
Time Frame: Baseline and Week 12
Population: Participants in safety population whose case report form contained baseline and Week 12 data for LDL-C levels.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 274
mg/dL | -6.81 (29.20)

5. Primary Outcome: Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Description: Serum HDL-C levels were measured at start of treatment (baseline) and after 12 weeks of treatment with TREDAPTIVE
Time Frame: Baseline and Week 12
Population: Participants in safety population whose case report form contained baseline and Week 12 data for HDL-C levels.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 294
mg/dL | 7.06 (9.53)

6. Primary Outcome: Change From Baseline in Triglycerides at Week 12
Description: Serum triglyceride levels were measured at start of treatment (baseline) and after 12 weeks of treatment with TREDAPTIVE
Time Frame: Baseline and Week 12
Population: Participants in safety population whose case report form contained baseline and Week 12 data for triglyceride levels.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 300
mg/dL | -106.32 (208.38)

7. Primary Outcome: Change From Baseline in Total Cholesterol at Week 24
Description: Serum cholesterol levels were measured at start of treatment (baseline) and after 24 weeks of treatment with TREDAPTIVE
Time Frame: Baseline and Week 24
Population: Participants in safety population whose case report form contained baseline and Week 24 data for total cholesterol levels and had received TREDAPTIVE for 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 76
mg/dL | -20.01 (35.08)

8. Primary Outcome: Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 24
Description: Serum LDL-C levels were measured at start of treatment (baseline) and after 24 weeks of treatment with TREDAPTIVE
Time Frame: Baseline and Week 24
Population: Participants in safety population whose case report form contained baseline and Week 24 data for LDL-C levels and had received TREDAPTIVE for 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 68
mg/dL | -14.82 (30.09)

9. Primary Outcome: Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 24
Description: Serum HDL-C levels were measured at start of treatment (baseline) and after 24 weeks of treatment with TREDAPTIVE
Time Frame: Baseline and Week 24
Population: Participants in safety population whose case report form contained baseline and Week 24 data for HDL-C levels and had received TREDAPTIVE for 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 72
mg/dL | 6.25 (8.70)

10. Primary Outcome: Change From Baseline in Triglycerides at Week 24
Description: Serum triglyceride levels were measured at start of treatment (baseline) and after 24 weeks of treatment with TREDAPTIVE
Time Frame: Baseline and Week 24
Population: Participants in safety population whose case report form contained baseline and Week 24 data for triglyceride levels and had received TREDAPTIVE for 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 75
mg/dL | -137.87 (153.24)

11. Primary Outcome: Investigator's Overall Efficacy Evaluation at Week 12
Description: The investigator evaluated all available data after 12 weeks of TREDAPTIVE and assigned an overall evaluation of "Improved", "Unchanged" or "Worsened" when compared to baseline.
Time Frame: Baseline and Week 12
Population: Participants in safety population whose case report form contained the investigator's overall assessment after 12 weeks of treatment with TREDAPTIVE
Measure: Number; unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 406
Percentage of Participants
  Improved | 68.23
  Unchanged | 25.86
  Worsened | 5.91

12. Primary Outcome: Investigator's Overall Efficacy Evaluation at Week 24
Description: The investigator evaluated all available data after 24 weeks of TREDAPTIVE and assigned an overall evaluation of "Improved", "Unchanged" or "Worsened" when compared to baseline.
Time Frame: Baseline and Week 24
Population: Participants in safety population whose case report form contained the investigator's overall assessment after 24 weeks of treatment with TREDAPTIVE
Measure: Number; unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 131
Percentage of Participants
  Improved | 72.52
  Unchanged | 20.61
  Worsened | 6.87

ADVERSE EVENTS:
Time Frame: From start of treatment through 14 days after the last dose (Up to 26 weeks)
Description: Safety population: all enrolled participants who met entry criteria regarding safety data
Arm/Group | ALL PARTICIPANTS
Serious Adverse Events (participants affected / at risk) | 7/862
Other Adverse Events (participants affected / at risk) | 65/862
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL PARTICIPANTS (N=862)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 3 (3)
UPPER EXTREMITY MASS (Musculoskeletal and connective tissue disorders) | 1 (1)
COMMUNICATION DISORDER (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL PARTICIPANTS (N=862)
PRURITUS (Skin and subcutaneous tissue disorders) | 65 (65)

LIMITATIONS AND CAVEATS:
Study enrollment stopped early due to termination of all TREDAPTIVE studies. Data obtained for participants enrolled prior to termination was analyzed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication must be approved by the Sponsor.